CLINICAL TRIAL: NCT01147497
Title: A Randomized Control Trial of Misoprostol Versus Placebo for Cervical Priming in Intrauterine Device Insertion for Nulliparous Women
Brief Title: Misoprostol Prior to Intrauterine Device (IUD) Insertion in Nulliparous Women
Acronym: miso
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Eva Lathrop, MD, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00021303; MISO Emory (Other: Other)
Record Dates: First submitted 2010-06-15; First posted 2010-06-22 (Estimated); Results first posted 2014-03-24 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Contraception
Keywords: IUD insertion; nulliparous women; contraception; family planning; IUD insertion in nulliparous women
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- misoprostol (Experimental): Misoprostol 400mcg taken buccally 2 hours prior to IUD insertion visit
  Interventions: Drug: Misoprostol
- placebo (Placebo Comparator): Pill that is identical to the study drug in appearance, taste, and smell, taken buccally 2 hours prior to IUD insertion visit
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol — 400mcg of misoprostol taken buccally 2 hours prior to IUD insertion visit
  Arms: misoprostol
Drug: Placebo — Pill that is identical to the study drug in appearance, taste and smell, taken buccally 2 hours prior to IUD insertion visit
  Arms: placebo

SUMMARY:
Because of misoprostol's known ability to cause cervical dilation, some family planning providers give their patients a dose of this drug prior to insertion. The goal of this study is to evaluate whether misoprostol prior to IUD insertion in nulliparous women eases insertion and decreases pain.

DETAILED DESCRIPTION:
There are currently 2 intrauterine devices (IUDs) available in the U.S., the copper T380 (paragard) and levonorgestrel IUD (Mirena). The effectiveness of IUDs is very similar to tubal sterilization[1], with an overall unintended pregnancy rate of less than 1% in the first year, and lower failure rates in subsequent years. The cervix of a nulliparous woman has a smaller diameter and can lead to more difficult and uncomfortable IUD insertions. Because of misoprostol's known ability to cause cervical dilation, some family planning providers give their patients a dose of this drug prior to insertion. The goal of this study is to evaluate whether misoprostol prior to IUD insertion in nulliparous women eases insertion and decreases pain. The null hypothesis is that misoprostol does not influence difficulty of insertion or patient perception of pain. The primary outcome is the ability to insert the IUD without dilation of the cervix or using ultrasound for guidance.

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* negative pregnancy test
* no prior pregnancy beyond 19 6/7 weeks
* no pelvic inflammatory disease in last 3 months
* no current cervicitis
* willing to follow up in 1-2 months

Exclusion Criteria:

* active cervical infection
* current pregnancy
* prior pregnancy beyond 19 6/7 weeks
* uterine anomaly
* fibroid uterus distorting uterine cavity
* copper allergy or wilson's disease for ParaGard
* undiagnosed abnormal uterine bleeding
* cervical or uterine cancer
* sepsis associated with the most recent pregnancy
* current breast cancer for levonogestrel IUD
* inflammatory bowel disease
* allergy to misoprostol

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Lathrop, MD, MPH, Principal Investigator — Emory University School of Medicine, Department of Gynecology and Obstetrics
Locations (1):
- The Emory Clinic, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Lathrop E, Haddad L, McWhorter CP, Goedken P. Self-administration of misoprostol prior to intrauterine device insertion among nulliparous women: a randomized controlled trial. Contraception. 2013 Dec;88(6):725-9. doi: 10.1016/j.contraception.2013.07.011. Epub 2013 Aug 6. PMID 24034580
- [Derived] Turok DK, Espey E, Edelman AB, Lotke PS, Lathrop EH, Teal SB, Jacobson JC, Simonsen SE, Schulz KF. The methodology for developing a prospective meta-analysis in the family planning community. Trials. 2011 Apr 29;12:104. doi: 10.1186/1745-6215-12-104. PMID 21527040

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred at a faculty practice clinic affiliated with Emory University.
Pre-assignment Details: Seventy-eight nulliparous women were enrolled, and 71 completed the study. Five dropped out prior to randomization and method insertion choosing other birth control options.
Period: Overall Study
Arm/Group | Misoprostol | Placebo
Started | 37 | 36
Completed | 35 | 36
Not Completed | 2 | 0
Not completed — failed insertion | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Misoprostol | Placebo | Total
Number analyzed (Participants) | 37 | 36 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 36 | 73
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.05 (.554) | 25.5 (.554) | 25.775 (.554)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 36 | 73
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 36 | 73

OUTCOME MEASURES:

1. Primary Outcome: Provider Perceived Ease of Insertion on a 100 Point Visual Analogue Scale
Description: The visual analogue scale for perceived ease ranges from 0 (most ease) to 100 (most difficult).
Time Frame: assessed immediately post IUD insertion
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Misoprostol | Placebo
Number analyzed (Participants) | 35 | 36
units on a scale | 21 [0 to 100] | 21 [0 to 68]

2. Secondary Outcome: Patient Perceived Pain on a 100 Point Visual Analogue Scale
Description: The visual analogue scale for perceived patient pain ranges from 0 (no pain) to 100 (most pain).
Time Frame: immediately after insertion
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Misoprostol | Placebo
Number analyzed (Participants) | 37 | 36
units on a scale | 46 [11 to 92] | 34 [0 to 90]

3. Secondary Outcome: The Use of Adjunctive Measures Including Ultrasound Guidance or Cervical Dilation to Insert the IUD
Time Frame: assessed immediately after IUD insertion
Measure: Number; unit: participants
Arm/Group | Misoprostol | Placebo
Number analyzed (Participants) | 37 | 36
participants | 7 | 3

4. Secondary Outcome: Time for Insertion Procedure
Time Frame: assessed immediately after IUD insertion
Population: Data were not collected for this outcome measure. The provider questionnaire developed for this study was piloted prior to study initiation and this question was removed for clarity and to focus on the primary study aims.
Arm/Group | Misoprostol | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Acceptability of Discomfort Associated With Insertion
Time Frame: assessed at one week after insertion and at one month after insertion
Population: Data were not collected for this outcome measure. The follow-up participant questionnaires developed for this study were piloted prior to study initiation and this question was removed for clarity, to focus on the primary study aims, and to reduce participant burden.
Arm/Group | Misoprostol | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Ease of Insertion and Presence of Pain in Nulliparous Women Versus Nulligravid Women
Time Frame: assessed immediately following insertion
Population: Data were not collected for this outcome measure. The participant questionnaire developed for this study was piloted prior to study initiation and some questions (including questions about prior pregnancies) were removed for clarity, to focus on the primary study aims, and to reduce participant burden.
Arm/Group | Misoprostol | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Need for Additional Pain Medications After Insertion of the IUD
Time Frame: assessed one week after insertion
Population: Data were not collected for this outcome measure. The follow-up questionnaire developed for this study was piloted prior to study initiation and some questions (including questions about medication use) were removed for clarity, to focus on the primary study aims, and to reduce participant burden.
Arm/Group | Misoprostol | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Misoprostol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/36
Other Adverse Events (participants affected / at risk) | 0/37 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No